CLINICAL TRIAL: NCT03603769
Title: In Vitro And Ex Vivo Anti-Inflammatory Activities Of Salmon Polar Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Responsible Party: Principal Investigator, Ioannis Zabetakis, Principal Investigator, University of Limerick
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: IP 2017 0518
Record Dates: First submitted 2017-12-07; First posted 2018-07-27 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Each subject will participate in five daily trials on 5 separate days, at least 2 weeks apart.
  Within each appointment each participant will come (after fasting overnight, 10-12 h), to our metabolic unit early in the morning (07:30 - 08.30 am) and will initially give a fasting baseline blood sample. Afterwards, in specific time he/she will be provided to consume a standardized breakfast and then he/she will be administered randomly either placebo or several versions of the food supplement containing Salmon Polar Lipids (Low Dose stomach release or High Dose stomach release or Low Dose intestine release or High Dose Intestine Release). Thus, the sequence of the trials will be randomly selected for each subject.
Who Masked: Participant, Investigator
Masking Description: A placebo capsule (glycerine only, with no SPL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Food Supplement (Salmon Polar Lipids) Intervention (Experimental): Experimental: After fasting overnight, subjects will come to our metabolic unit where in a randomized and double blinded way they will be provided several versions of the food supplement either of stomach resistant (intestine release) or stomach non-resistant (stomach release) each containing either 0.25 (Low Dose) or 0.50 g (High Dose) of Salmon Polar Lipids (SPL)
  Assessment & outcome measured: Blood samples will be taken from each subject at baseline (0 hours) and after 1-4 hours of the SPL-food supplement intervention. Aggregation of platelets will be assessed in these samples as previously described (see references 1-4), in order to evaluate the postprandial effects of this supplement on platelet aggregation.
  Other blood coagulation parameters will also be evaluated, such as prothrombin time, fibrinogen, Activated partial thromboplastin time Plasma lipid profile (levels of plasma Total Cholesterol, LDL, HDL and Triglycerides) and serum CRP levels will also be assessed.
  Interventions: Dietary Supplement: Food supplement capsules containing Salmon-Polar Lipids
- Group B: Consumption of Placebo Comparator (Placebo Comparator): Experimental: After fasting overnight subjects will come to the metabolic unit in UL at 08.00 am where in a randomized and double blinded way they will be provided a placebo capsule containing only glycerin.
  Assessment & outcome measured: Blood samples will be taken from each subject at baseline (0 hours) and after 1-4 hours of the placebo administration. Aggregation of their platelets will be assessed as previously described (see references 1-4), in order to evaluate the postprandial effects of this supplement on platelet aggregation.
  Other blood coagulation parameters will also be evaluated, such as prothrombin time, fibrinogen, Activated partial thromboplastin time Plasma lipid profile (levels of plasma Total Cholesterol, LDL, HDL and Triglycerides) and serum CRP levels will also be assessed.
  Interventions: Dietary Supplement: Placebo food supplement capsule

INTERVENTIONS:
Dietary Supplement: Food supplement capsules containing Salmon-Polar Lipids — Postprandial decreased Platelet activation/aggregation in subjects, after the food supplement capsule consumption
  Arms: Group A: Food Supplement (Salmon Polar Lipids) Intervention
Dietary Supplement: Placebo food supplement capsule — Postprandial unaffected platelet activation/aggregation in subjects, after the food supplement capsule consumption
  Arms: Group B: Consumption of Placebo Comparator

SUMMARY:
The aim of this project is to study the effects of a new-developed food-supplement that contains bioactive polar lipids derived from organic farmed Irish salmon for the beneficial promotion of cardiovascular health. The health claims that will be formulated for this nutraceutical are based on EFSA guidelines "The scientific requirements for health claims related to antioxidants, oxidative damage and cardiovascular health" and in particular paragraph 5.4, "Claims on reduced platelet aggregation" "Platelet hyperactivity and hypercoagulability states are more commonly observed in subjects with cardiovascular (CV) risk factors. Healthy subjects at very low risk of CV disease normally have non-activated circulating platelets. Decreasing platelet aggregation in subjects with platelet activation during sustained exposure to the food/constituent (e.g. four weeks) would be a beneficial physiological effect".

Within this study, the postprandial effects of this novel food supplement against platelet aggregation and inflammation are going to be exploited ex vivo in blood from human subjects as described in previously established procedures.

ELIGIBILITY:
Inclusion Criteria:

Subjects need to:

* Have their dietary intake of fish to be within normal range (1-2 portions per week).

Exclusion Criteria:

Subjects will be excluded if they:

* Are currently taking medication and/or dietary supplements
* Have blood clotting disorders or dislipidemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Postprandial effect of Supplement/placebo on human platelet aggregation induced by Platelet Activating Factor (PAF) | 2 Months
  Bio-assays on platelets will be assessed as previously described. Briefly:
  Standard PAF dissolved in BSA will have final concentrations 2.6e-8 - 2.6e-5 mol/L when testing into a Chronolog-490 two channel turbidimetric platelet aggregometer. The maximum reversible or the minimum irreversible PAF-induced platelet aggregation is determined as the 100% aggregation, and then various PAF concentrations are added, so as to achieve aggregations between 20% and 80% aggregation, which are of linear response to the added PAF concentration. The EC50 value that accounts for the PAF concentration (mol/L) inducing 50% aggregation of human platelets will be calculated by the equation derived from this linear curve. Results will be expressed as percentage change of EC50 on 1, 2, 3 and 4 hours of the food supplement/placebo administration, compared with baseline (0 hours)

SECONDARY OUTCOMES:
Postprandial effect of Supplement/placebo on human platelet aggregation induced by Thrombin | 2 Months
  Bio-assays on platelets will be assessed as previously described. Briefly:
  Standard active thrombin dissolved in saline will have final concentrations 0.01 - 1.0 IU/mL when testing into a Chronolog-490 two channel turbidimetric platelet aggregometer. The maximum reversible or the minimum irreversible Thrombin-induced platelet aggregation is determined as the 100% aggregation, and then various Thrombin concentrations are added, so as to achieve aggregations between 20% and 80% aggregation, which are of linear response to the added Thrombin concentration. The EC50 value that accounts for the Thrombin concentration (IU/mL) inducing 50% aggregation of human platelets will be calculated by the equation derived from this linear curve. Results will be expressed as percentage change of EC50 on 1, 2, 3 and 4 hours of the food supplement/placebo administration, compared with baseline (0 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Zabetakis, Dr, Principal Investigator — University of Limerick
Locations (1):
- Department of Biological Sciences, Limerick, Co. Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsoupras A, Lordan R, Demuru M, Shiels K, Saha SK, Nasopoulou C, Zabetakis I. Structural Elucidation of Irish Organic Farmed Salmon (Salmo salar) Polar Lipids with Antithrombotic Activities. Mar Drugs. 2018 May 23;16(6):176. doi: 10.3390/md16060176. PMID 29882848
- [Background] Nasopoulou C, Tsoupras AB, Karantonis HC, Demopoulos CA, Zabetakis I. Fish polar lipids retard atherosclerosis in rabbits by down-regulating PAF biosynthesis and up-regulating PAF catabolism. Lipids Health Dis. 2011 Nov 16;10:213. doi: 10.1186/1476-511X-10-213. PMID 22087726
- [Background] Tsantila N, Tsoupras AB, Fragopoulou E, Antonopoulou S, Iatrou C, Demopoulos CA. In vitro and in vivo effects of statins on platelet-activating factor and its metabolism. Angiology. 2011 Apr;62(3):209-18. doi: 10.1177/0003319710375089. Epub 2010 Aug 29. PMID 20805097
- [Background] Xanthopoulou MN, Kalathara K, Melachroinou S, Arampatzi-Menenakou K, Antonopoulou S, Yannakoulia M, Fragopoulou E. Wine consumption reduced postprandial platelet sensitivity against platelet activating factor in healthy men. Eur J Nutr. 2017 Jun;56(4):1485-1492. doi: 10.1007/s00394-016-1194-0. Epub 2016 Mar 2. PMID 26936842